CLINICAL TRIAL: NCT06092814
Title: Transcranial Alternating Current Stimulation (tACS) to Enhance Language Abilities
Brief Title: tACS to Enhance Language Abilities
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 854139
Record Dates: First submitted 2023-09-28; First posted 2023-10-23 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Aphasia, Acquired; Aphasia
Keywords: non-invasive brain stimulation; transcranial alternating current stimulation (tACS); EEG
MeSH Terms: conditions — Stroke; Aphasia

STUDY DESIGN:
Intervention Model Description: The proposed study is a within-subject, double-blind & sham-controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real-tACS (Active Comparator): The active stimulation will consist of an alternating current delivered in the alpha frequency band with a peak-to-peak intensity of 4 milliamps (mA) for 20 minutes. Participants will complete sentence completion and verb generation task during stimulation.
  Interventions: Device: Active transcranial alternating current stimulation (tACS)
- sham-tACS (Placebo Comparator): Sham stimulation involves the delivery of 60 seconds of the actual stimulation waveform ("ramp up") which is then gradually reduced to 0 milliamps (mA) ("ramp down"). Participants will complete sentence completion and verb generation task during stimulation.
  Interventions: Device: Active transcranial alternating current stimulation (tACS)

INTERVENTIONS:
Device: Active transcranial alternating current stimulation (tACS) — Transcranial Alternating Current Stimulation (tACS) is a device that applies a low-intensity electrical current to the brain through electrodes on the scalp.
  Other Names: Sham transcranial alternating current stimulation [(ACS)

SUMMARY:
The goal of this study is to see if transcranial alternating current stimulation (tACS) can be used to enhance language abilities in people with post-stroke aphasia. Participants will receive real and sham tACS in conjunction with various language tests. Researchers will compare the post-stroke aphasia group with aged matched controls to see if brain response to tACS differs between groups.

DETAILED DESCRIPTION:
This research will investigate whether transcranial alternating current stimulation (tACS), a form of noninvasive brain stimulation, can be used to enhance language abilities in people with aphasia (PWA) due to stroke and healthy older adults when compared to placebo (sham) tACS. The investigators hypothesize that alpha vs. sham tACS will improve language abilities. In addition, the investigators propose that alpha vs. sham tACS will increase local alpha power as well as alpha-induced functional connectivity, and the degree to which alpha tACS increases will be related to the degree of language performance improvement. Finally, the investigators hypothesize that PWA will exhibit abnormalities in alpha-related activity when compared to matched controls, and aphasia severity will be associated with the degree of PWA dysfunction in alpha power and alpha-driven functional connectivity.

ELIGIBILITY:
Inclusion Criteria for Persons with Aphasia:

1. Presence of aphasia
2. Suffered a single, left hemisphere stroke
3. Stroke ≥6 months old (chronic) at the time of enrollment

Inclusion Criteria for Healthy Controls:

1. Right-handedness
2. Must be able to understand the nature of the study, and give informed consent

Exclusion criteria for Persons with Aphasia:

1. Inability to understand the nature of the study
2. Marked naming impairment
3. Impaired non-verbal, conceptual processing
4. History of significant medical or neurological disorder (other than stroke)
5. History of significant or poorly controlled psychiatric disorders
6. Current abuse of alcohol or drugs, prescription or otherwise
7. Nursing a child, pregnancy, or intent to become pregnant during the study
8. Clinically significant hearing loss
9. Contraindications to tACS
10. Contraindications to MRI

Exclusion Criteria for Healthy Controls

1. Diagnosis of a neurodegenerative disease or clinically significant cognitive complaint
2. Any unrelated neurologic or physical condition that impairs communication ability
3. History of unrelated neurological conditions including but not limited to traumatic brain injury, stroke, or small vessel disease that has resulted in a neurologic deficit
4. Any additional neurological condition that would likely reduce the safety of study participation, including central nervous system (CNS) vasculitis, intracranial tumor, intracranial aneurysm, multiple sclerosis or arteriovenous malformations
5. A medically unstable cardiopulmonary or metabolic disorder
6. Terminal illness associated with survival <12 months
7. Major active psychiatric illness that may interfere with required study procedures or treatments as determined by the enrolling physician
8. Current abuse of alcohol or drugs, prescription or otherwise
9. Contraindications to tACS
10. Contraindications to MRI

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-12 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Performance on the Blocked-Cyclic Naming (BCN) Task | 5-10 minutes after a single session of active (alpha tACS) and sham (fake tACS).
  The BCN tasks involves naming a set of pictures repeatedly. Sets of pictures come from either the same semantic category (high competition condition; e.g., categorically related: "dog", "cat", "panda") or different semantic categories (low competition condition; e.g., unrelated: dog, eye, crib).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States